CLINICAL TRIAL: NCT03683238
Title: Role of Nutritionist in the Multidisciplinary Approach of Hidradenitis Suppurativa (Acne Inversa)
Brief Title: Nutritional Status and Hidradenitis Suppurativa (Acne Inversa)
Acronym: NutriHidra
Status: Completed | Type: Observational
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Prof. Silvia Savastano, Associate Professor, Federico II University
Other Study IDs: 201/15
Record Dates: First submitted 2018-07-10; First posted 2018-09-25 (Actual); Last update posted 2018-09-25 (Actual); Status verified 2018-09

CONDITIONS: Hidradenitis Suppurativa; Mediterranean Diet; Body Composition; Vitamin D Deficiency; Trimethylamine N-oxide (TMAO)
MeSH Terms: conditions — Hidradenitis Suppurativa; Vitamin D Deficiency | interventions — Diet, Mediterranean

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Dietary Supplement: Mediterranean Diet — We aim to determine the effects of the traditional Mediterranean Diet on Hidradenitis suppurativa

SUMMARY:
Hidradenitis suppurativa (HS) is a chronic inflammatory, debilitating skin disorder. The exacerbating factors of HS include nutrition and adiposity. The objective of this study was to investigate the relationships between body composition and the adherence to the Mediterranean diet (MD) with the severity of HS in a sample of naïve-treatment patients with HS. In the wake of this evidence, in the study to investigate the relationships between nutritional status, the adherence to the MD, body composition, and the severity of HS in a sample of naïve-treatment patients with HS compared to control group matched for sex, age, and body weight.

ELIGIBILITY:
Inclusion Criteria:

* healthy subjects of both gender
* treatment-naïve patients
* had HS diagnosed ≥6 months before study initiation wash out therapy for at least 3 months

Exclusion Criteria:

* occasional or current of use of drugs for HS, including topical antibiotics and systemic treatments (such as clindamycin-rifampicin, tetracycline, Rifampicin-moxifloxacin-metronidazole, ertapenem, acitretin, cyclosporine A, dapsone, isotretinoin, biologics;
* hypocaloric diet in the last three months or specific nutritional regimens;
* vitamin/mineral or antioxidant supplementation;
* occasional or current of use of drugs that could influence fluid balance, including non-steroidal anti-inflammatory drugs, hormone replacement therapy.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Study population consisted of 82 participants, 41 patients with HS and 41 healthy subjects as control group.
Sampling Method: Non-Probability Sample
Enrollment: 81 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2018-04 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
Adherence to Mediterranean Diet by Predimed Questionnaire | April 2015 to April 2018
  Validated 14-item tool of adherence to the Mediterranean diet, with three categories of adherence (≤5, low adherence, 6-9, average adherence and ≥10 points, high adherence)
Phase angle | April 2015 to April 2018
  Phase angle was performed using a BIA phase-sensitive system by experienced observers (an 800-µA current at a frequency single-frequency of 50 kHz BIA 101 RJL, Akern Bioresearch, Florence, Italy).
Trimethylamine N-oxide plasma levels | April 2015 to April 2018
  ultra high-performance liquid chromatography

SECONDARY OUTCOMES:
Vitamin D | April 2015 to April 2018
  25 OH vitamin D assay for the LIAISON automated analyzer

IPD SHARING:
Plan to Share IPD: No